CLINICAL TRIAL: NCT05414474
Title: Effects of Nutritional Iron Absorption Enhancers and Inhibitors and Daytime on Absorption From Oral Iron Supplements
Brief Title: Effects of Enhancers and Inhibitors on Absorption From Iron Supplements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IDEA
Record Dates: First submitted 2022-05-13; First posted 2022-06-10 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Iron-deficiency; Iron Deficiency Anemia
Keywords: iron supplementation; women of reproductive age; iron absorption enhancers; iron absorption inhibitors; ferrous fumarate; iron deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency; Iron Deficiencies | interventions — Ascorbic Acid; Coffee; Breakfast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Reference (Active Comparator): Ferrum Hausmann 100 mg is consumed with 200 mL nanopure water with labelled ferrous fumarate (3 mg 54Fe).
  Interventions: Other: Reference
- Ascorbic acid (AA) 500 mg (Experimental): Ferrum Hausmann 100 mg is consumed with 200 mL nanopure water with labelled ferrous fumarate (3 mg 57Fe) and 500 mg AA.
  Interventions: Other: Ascorbic acid (AA) 500 mg
- Ascorbic acid (AA) 80 mg (Experimental): Ferrum Hausmann 100 mg is consumed with 200 mL nanopure water with labelled ferrous fumarate (3 mg 58Fe) and 80 mg AA.
  Interventions: Other: Ascorbic acid (AA) 80 mg
- Coffee (Experimental): Ferrum Hausmann 100 mg is consumed with 200 mL nanopure water with labelled ferrous fumarate (3 mg 54Fe) and 150 mL coffee.
  Interventions: Other: Coffee
- Breakfast (Experimental): Ferrum Hausmann 100 mg is consumed with 200 mL nanopure water with labelled ferrous fumarate (3 mg 57Fe) and 1 bread roll (~100 g) with butter and honey, 1 cup of plain yoghurt (180 mL), 1 cup of coffee (150 mL) and 1 glass of orange juice (250 mL).
  Interventions: Other: Breakfast
- Afternoon (Experimental): Ferrum Hausmann 100 mg is consumed with 200 mL nanopure water with labelled ferrous fumarate (3 mg 58Fe) in the afternoon .
  Interventions: Other: Afternoon

INTERVENTIONS:
Other: Reference — Ferrum Hausmann 100 mg + 200 mL nanopure water with 3 mg 54Fe isotopes
  Arms: Reference
Other: Ascorbic acid (AA) 500 mg — Ferrum Hausmann 100 mg + 200 mL nanopure water with 3 mg 57Fe isotopes + 500 mg AA
  Arms: Ascorbic acid (AA) 500 mg
Other: Ascorbic acid (AA) 80 mg — Ferrum Hausmann 100 mg + 200 mL nanopure water with 3 mg 58Fe + 80 mg AA
  Arms: Ascorbic acid (AA) 80 mg
Other: Coffee — Ferrum Hausmann 100 mg + 200 mL nanopure water with 3 mg 54Fe isotopes + 150 mL coffee
  Arms: Coffee
Other: Breakfast — Ferrum Hausmann 100 mg + 200 mL nanopure water with 3 mg 57Fe isotopes + 1 bread roll (~100 g) with butter and honey + 1 cup of plain yoghurt (180 mL) + 1 cup of coffee (150 mL) + 1 glass of orange juice (250 mL)
  Arms: Breakfast
Other: Afternoon — Ferrum Hausmann 100 mg + 200 mL nanopure water with 3 mg 58Fe isotopes administered in the afternoon
  Arms: Afternoon

SUMMARY:
Iron deficiency (ID) is a major public health problem worldwide and oral iron supplementation can be an effective strategy to treat and prevent ID. To maximize iron bioavailability form oral iron supplements the simultaneous intake of the iron absorption enhancer ascorbic acid (AA) is recommended, and the simultaneous intake of coffee or tea containing the iron absorption inhibitors polyphenols should be avoided. Also, oral iron supplements are recommended to be taken on an empty stomach in the morning and without a meal to avoid any interaction with phytic acid, another iron absorption inhibitor present in many foods. However, the effects of these iron absorption enhancers and inhibitors have only been shown on iron absorption from dietary iron (up to 10mg). Also, the effect of the diurnal hepcidin increase on absorption from an iron supplement given in the afternoon without a preceding morning dose is unclear. Whether AA also increases iron bioavailability from a supplemental iron dose and whether a cup of coffee, a breakfast or iron administration in the afternoon decreases iron bioavailability from a supplemental dose is uncertain.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 to 45 years old,
* SF levels <30 μg/L,
* Body weight < 70 kg
* Normal Body Mass Index (18.5-25 kg/m2),
* Signed informed consent.

Exclusion Criteria:

* Anemia (Hb < 12 g/dL)
* Elevated CRP > 5 mg/L,
* Any metabolic, gastrointestinal, kidney or chronic disease such as diabetes, renal failure, hepatic dysfunction, hepatitis, hypertension, cancer or cardiovascular diseases (according to the participants own statement) affecting iron metabolism,
* Continuous/long-term use of medication during the whole study, which may interfere with iron absorption, gut physiology and iron metabolism,
* Consumption of mineral and vitamin supplements since screening and over the study period until last blood sample collection,
* Difficulties with blood sampling,
* Blood transfusion, blood donation or significant blood loss (accident, surgery) over the past 6 months,
* Known hypersensitivity or allergy to iron capsules in the given amount (ferrous fumarate, brilliant blue FCF (E133), titandioxide (E171) and sodium lauryl sulfate)
* Pregnancy, breastfeeding
* Women who intend to become pregnant during the course of the study,
* Known or suspected non-compliance, drug or alcohol (more than 2 drinks/day) abuse,
* Smokers (> 1 cigarette per week),
* Participant is likely to be absent on one the study appointments,
* Inability to follow the procedures of the study, e.g. due to language problems, self-reported psychological disorders, etc. of the participant.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
Fractional iron absorption [percent] | Day 22
  Fractional iron absorption will be calculated based on the shift of the iron isotope ratios in the collected blood samples after the administration of the intervention products. Fractional iron absorption will be measured as erythrocyte incorporation of the naturally occurring iron forms with different masses used to label the iron supplements.
Fractional iron absorption [percent] | Day 43
  Fractional iron absorption will be calculated based on the shift of the iron isotope ratios in the collected blood samples after the administration of the intervention products. Fractional iron absorption will be measured as erythrocyte incorporation of the naturally occurring iron forms with different masses used to label the iron supplements.
Total iron absorption [mg] | Day 22
  Total iron absorption will be calculated based on the shift of the iron isotope ratios in the collected blood samples after the administration of the intervention products. Total iron absorption will be measured as erythrocyte incorporation of the naturally occurring iron forms with different masses used to label the iron supplements.
Total iron absorption [mg] | Day 43
  Total iron absorption will be calculated based on the shift of the iron isotope ratios in the collected blood samples after the administration of the intervention products. Total iron absorption will be measured as erythrocyte incorporation of the naturally occurring iron forms with different masses used to label the iron supplements.

SECONDARY OUTCOMES:
Hemoglobin (Hb) | Day 1, 22, 26 and 43
  Iron status marker
Serum ferritin (SF) | Day 1, 22, 26 and 43
  Iron status marker
Serum transferrin receptor (sTfR) | Day 1, 22, 26 and 43
  Iron status marker
Serum iron (SFe) | Day 1, 22, 26 and 43
  Iron status marker
Total iron binding capacity (TIBC) | Day 1, 22, 26 and 43
  Iron status marker
Hepcidin | Day 1, 22 and 26
  Iron regulatory protein
C-reactive protein (CRP) | Day 1, 22, 26 and 43
  Inflammation marker
Alpha-1-acid-glycoprotein (AGP) | Day 1, 22, 26 and 43
  Inflammation marker

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Stoffel, Dr., Principal Investigator — Human Nutrition Laboratory, ETH Zuerich
Locations (1):
- ETH Zurich; Human Nutrition Laboratory; Institute of Food, Nutrition and Health, Zurich, Switzerland